CLINICAL TRIAL: NCT03919474
Title: Markers of Microvascular Lesion in Adult Patients With Acquired Sudden Cochelo-vestibular Deficiency
Brief Title: Blood Markers in Adult Patients With Sudden Sensorineural Hearing Loss (SSNHL)
Acronym: SSNHL
Status: Completed | Type: Observational
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Ludovic Drouet MD, PhD, Principal Investigator, Hopital Lariboisière
Other Study IDs: HLariboisiere-ORL
Record Dates: First submitted 2019-04-02; First posted 2019-04-18 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Idiopathic SSNHL; Age Over 18
Keywords: sudden hearing loss,; SSNHL; serotonin; homocystein; antiphospholipid syndrom; thrombophilia
MeSH Terms: conditions — Hearing Loss, Sudden; Thrombophilia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — venous peripheral blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: microvascular markers — follow up of microvascular biomarkers during patient follow up

SUMMARY:
The roles of thrombophilia and cardiovascular risk factors in sudden sensorineural hearing loss (SSNHL) remain controversial. Cochlear micro-thrombosis has been hypothesized as a possible pathogenic mechanism of SSNHL. The objective was thus to measure the levels of markers of macrovascular thrombosis and microvascular risk factors

DETAILED DESCRIPTION:
To recruit adult consecutive outpatients referred for SSNHL to the otolaryngologist clinic of our university hospital starting June 2016 and prospectively until december 31th 2018.

Plasma sampling and biomarkers quantification : After a 48-hours diet excluding serotonin- and tryptophan-rich food, fasting blood samples were collected into vacuum tubes containing 109 mM sodium citrate (Becton-Dickinson, Le Pont de Claix, France) with a 9:1 blood-to-anticoagulant ratio. After removing 0.5 mL of whole blood for serotonin measurements, the remainder was centrifuged at 1,000 x g for 10 minutes, and the supernatant was then centrifuged at 3,000 x g for 15 minutes to isolate platelets and obtain platelet-poor plasma. Importantly, the time between blood sampling and platelet/plasma isolation was less than one hour. Aliquots of whole blood, platelets, and plasma were kept frozen (-20°C) until serotonin and homocysteine measurements performed within one week after congelation. Whole blood, platelet and plasma 5-HT as well as plasma homocysteine (Hcy) levels were measured by high pressure liquid chromatography coupled to fluorimetric detections .

Thrombophilia screening included measurements of antithrombin , protein C, protein S, factor V Leiden, prothrombin G20210A, methylene tetrahydrofolate reductase (MTHFR) C677T, antiphospholipid antibodies anticardiolipin IgG and IgM and anti-beta2 glycoprotein 1 IgG), dilute Russell viper venom time , Rosner index, factor VIII, von Willebrand factor (vWF) activity and antigen. Tests were performed on citrated plasma, serum or DNA as appropriate and as previously described

ELIGIBILITY:
Inclusion Criteria:

* adult idiopathic SSNHL

Exclusion Criteria:

* secundary hearing loss

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: unrelated adult consecutive outpatients referred for SSNHL to the otolaryngologist clinic of our university hospital
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
change from Baseline of plasma serotonin at three months | at three months and then once a year up to five years
  plasma serotonin level (HPLC, frequent value <15nM)
change from Baseline of plasma homocystein at three months | at three months and then once a year up to five years
  plasma homocystein (HPLC, fequent value <15 µM)
change from Baseline serum of anticardiolipine antibody at three months | at three months and then once a year up to five years
  serum anticardiolipin antiboy (ELISA, frequent value <10units)

SECONDARY OUTCOMES:
change from Baseline of hearing characteristics at three months | at three months and then once a year up to five years
  audiogram

CONTACTS AND LOCATIONS:
Overall Officials: jean-marie Launay, PharmD, PhD, Study Director — Hopital Lariboisière
Locations (1):
- HLariboisier otholaryngology clinic, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided
it will be decided at completion of patient recruitement

REFERENCES:
- [Background] Callebert J, Esteve JM, Herve P, Peoc'h K, Tournois C, Drouet L, Launay JM, Maroteaux L. Evidence for a control of plasma serotonin levels by 5-hydroxytryptamine(2B) receptors in mice. J Pharmacol Exp Ther. 2006 May;317(2):724-31. doi: 10.1124/jpet.105.098269. Epub 2006 Feb 3. PMID 16461587
- [Result] Brand T, Anderson GM. The measurement of platelet-poor plasma serotonin: a systematic review of prior reports and recommendations for improved analysis. Clin Chem. 2011 Oct;57(10):1376-86. doi: 10.1373/clinchem.2011.163824. Epub 2011 Aug 22. PMID 21859903